CLINICAL TRIAL: NCT03187405
Title: Intraventricular Fibrinolysis Versus External Ventricular Drainage Alone in Aneurysmal Subarachnoid Hemorrhage: a Randomized Controlled Trial.
Brief Title: Intraventricular Fibrinolysis for Aneurysmal Subarachnoid Hemorrhage.
Acronym: FIVHeMA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of patient
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIVHeMA
Record Dates: First submitted 2017-06-06; First posted 2017-06-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Hemorrhage; Intracranial Aneurysm; Cerebral Ischemia; Ventriculostomy; Tissue Plasminogen Activator
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm; Brain Ischemia | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: We plan to perform a pragmatic randomized controlled trial: compare the standard of care, i.e. the EVD alone, to the experimental treatment, i.e. IVF. As the standard treatment does not include injection within the EVD, the trial will not include injection through the EVD in the control group, so the trial will have an open design.
Who Masked: Outcomes Assessor
Masking Description: To minimize bias, the randomization and the treatment from V0 to the end of treatment will be performed by the local intensivist designed as investigator. The follow-up until day 4 (V1) to 6 months (V4), so the judgement criteria will be collected by the local neurosurgeon designed as investigator, who will be blinded to the treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVD alone (No Intervention): In the EVD alone group group, the EVD will be managed as usual - i.e. will only be used to drain CSF.
- EVD + IVF with Alteplase (Experimental): Intraventricular fibrinolysis: Injection through the EVD of 1mg in 1 mL of Alteplase every eight hours during 3 days (9 doses).
  Interventions: Drug: EVD + IVF with Alteplase

INTERVENTIONS:
Drug: EVD + IVF with Alteplase — Intraventricular fibrinolysis: Injection through the EVD of 1mg in 1 mL of Alteplase every eight hours during 3 days (9 doses).
  Other Names: Intraventricular fibrinolysis with Alteplase
  Arms: EVD + IVF with Alteplase

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) is a devastating form of stroke, with delayed cerebral ischemia (DCI) as a major complication. There are several evidences, both in preclinical and in clinical studies that intraventricular fibrinolysis (IVF) controls the phenomenon that are leading to DCI. Here, the investigators propose to conduct a phase III trial to provide a clear evaluation of the impact of IVF after aneurysmal SAH.

DETAILED DESCRIPTION:
Introduction: Aneurysmal subarachnoid hemorrhage (SAH) is a devastating form of stroke, which often causes acute hydrocephalus requiring the insertion of an external ventricular drain (EVD). A major complication of aneurysmal SAH is delayed cerebral ischemia (DCI), which corresponds to the occurrence of an ischemic stroke up to 21 days after the aneurysm rupture. There are currently only few ways to prevent it. As DCI is linked to the presence of blood within the subarachnoid space, it has been hypothesized that removing this blood may decrease the risk of DCI. It could be obtained by injecting a fibrinolytic agent through the EVD, a therapeutic strategy named intraventricular fibrinolysis (IVF). There are several evidences, both in preclinical and in clinical studies that IVF controls the phenomenon that are leading to DCI. It has notably been shown in Phase I and Phase II trial that IVF in aneurysmal SAH is safe and may decrease the risk of DCI, with a trend to improve the rate of good functional outcome by about 10%. Here, the investigators propose to conduct a phase III trial to provide a clear evaluation of the impact of IVF after aneurysmal SAH.

Materials and methods: this study will include patients with aneurysmal SAH requiring external ventricular drainage. The investigators will perform a pragmatic randomized controlled trial: compare the standard of care, i.e. the EVD alone, to the experimental treatment, i.e. IVF, with an open design. After exclusion of the aneurysm, patients will be randomly allocated to receive either EVD alone or EVD+IVF (72 hours, 9 doses). The primary outcome will be the proportion of patients without severe disability 6 months after the aneurysm rupture, as evaluated by the modified Rankin Scale (mRS). The investigators plan to include 440 patients, to show an increase of the rate of good functional outcome of 10% in the EVD+IVF group compared to the EVD alone group (α=0.05 and β=0.8). To obtain such sample, a multicenter trial is mandatory, and to date 16 centers accepted to participate. Each center will include one patient per month, and the inclusion period is to last 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 18-75) with SAH on initial CT-Scan examination.
* SAH associated with hydrocephalus requiring external ventricular drainage.
* Confirmation of an associated intracranial aneurysm by vascular imaging.
* Time from onset to admission under 24 hours.
* Exclusion of the aneurysm by surgical clipping or endovascular coiling before IVF.
* Oral information on research and informed consent of the patient and/or his relatives.

Exclusion Criteria:

* Patient with severe clinical presentation on admission: WFNS score = 5.
* Associated intracerebral hematoma of more than 2 cm in its larger width.
* SAH diagnosed on lumbar puncture: original Fisher grade = 1.
* Impossibility to exclude the aneurysm within 72 hours following its rupture.
* Patient previously treated with antiplatelet therapy or treated with antiplatelet therapy after the aneurysm exclusion.
* Severe coagulopathy, including oral vitamin K antagonist.
* Pregnant or lactating woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Participants With Modified Rankin Scale (mRS) <=3 - Dichotomized Analysis. | 6 months.
  Proportion of patients without severe disability evaluated by the modified Rankin Scale (0-3). The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 (perfect health without symptoms) to 6 (death).

SECONDARY OUTCOMES:
Death | 6 months
  Risk of death
DCI. | 6 weeks
  The presence of cerebral infarction on CT or MR scan on the latest CT or MR scan made before death within 6 weeks, not present on the CT or MR scan between 24 and 48 hours after early aneurysm occlusion, and not attributable to other causes such as surgical clipping or endovascular treatment.
Clinical deterioration caused by DCI. | 1 month
  Occurrence of focal neurological impairment (such as hemiparesis, aphasia, apraxia, hemianopia, or neglect), or a decrease of at least 2 points on the Glasgow Coma Scale. This should last for at least 1 hour, is not apparent immediately after aneurysm occlusion, and cannot be attributed to other causes by means of clinical assessment, CT or MRI scanning of the brain, and appropriate laboratory studies
EVD obstruction. | 1 month
  Numbers of permanent catheter obstruction requiring the insertion of a new catheter.
Internal CSF shunt surgery. | 3 months
  Rate of internal CSF shunt surgery.
Rebleeding. | 4 days
  A new ICH identified on a CT-scan performed after IVF that was not present before IVF.
Catheter related infection. | 3 month
  Clinical picture of infection associated with a positive CSF culture.
Rate of patients who returned to work. | 6 months
  Proportion of patient who returned to their previous professional activity.
Quality of life evaluated by the MOS SF-36 scale | 6 months
  MOS SF-36 scale
Asthenia. | 6 months
  Asthenia scale of Pichot

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gaberel, MD, PhD, Study Chair — University Hospital, Caen
Locations (1):
- University Hospital Of Caen, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Etminan N, Beseoglu K, Eicker SO, Turowski B, Steiger HJ, Hanggi D. Prospective, randomized, open-label phase II trial on concomitant intraventricular fibrinolysis and low-frequency rotation after severe subarachnoid hemorrhage. Stroke. 2013 Aug;44(8):2162-8. doi: 10.1161/STROKEAHA.113.001790. Epub 2013 Jun 4. PMID 23735957
- [Background] Goulay R, Flament J, Gauberti M, Naveau M, Pasquet N, Gakuba C, Emery E, Hantraye P, Vivien D, Aron-Badin R, Gaberel T. Subarachnoid Hemorrhage Severely Impairs Brain Parenchymal Cerebrospinal Fluid Circulation in Nonhuman Primate. Stroke. 2017 Aug;48(8):2301-2305. doi: 10.1161/STROKEAHA.117.017014. Epub 2017 May 19. PMID 28526764
- [Background] Hanley DF, Lane K, McBee N, Ziai W, Tuhrim S, Lees KR, Dawson J, Gandhi D, Ullman N, Mould WA, Mayo SW, Mendelow AD, Gregson B, Butcher K, Vespa P, Wright DW, Kase CS, Carhuapoma JR, Keyl PM, Diener-West M, Muschelli J, Betz JF, Thompson CB, Sugar EA, Yenokyan G, Janis S, John S, Harnof S, Lopez GA, Aldrich EF, Harrigan MR, Ansari S, Jallo J, Caron JL, LeDoux D, Adeoye O, Zuccarello M, Adams HP Jr, Rosenblum M, Thompson RE, Awad IA; CLEAR III Investigators. Thrombolytic removal of intraventricular haemorrhage in treatment of severe stroke: results of the randomised, multicentre, multiregion, placebo-controlled CLEAR III trial. Lancet. 2017 Feb 11;389(10069):603-611. doi: 10.1016/S0140-6736(16)32410-2. Epub 2017 Jan 10. PMID 28081952